CLINICAL TRIAL: NCT05688956
Title: Protein Supplement and Exercise Training for the Treatment of Sarcopenia Risk in Older Adults Who Receive Supportive Home Care: POWER Study
Brief Title: Protein Supplement and Exercise Training for the Treatment of Sarcopenia Risk in Older Adults
Acronym: POWER
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University College Dublin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 107102
Record Dates: First submitted 2022-12-14; First posted 2023-01-18 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Sarcopenia
Keywords: Older adults; Home care; Community-dwelling; Sarcopenia; Oral Nutritional Supplement; Resistance exercise
MeSH Terms: conditions — Sarcopenia | interventions — Nutrition Assessment

STUDY DESIGN:
Intervention Model Description: A randomised, parallel group, 12-week clinical trial with two groups of older adults aged 70+ years requiring supportive home care will be undertaken.
Who Masked: Participant
Masking Description: Participants will be randomly assigned to either consume the oral nutritional supplement or not.
  Each participant will know if they are either taking the oral nutritional supplement or not. There is no placebo, ONS being provided. Standard dietary advice to increase intake of protein, leucine and vitamin D using available literature designed for those at risk of malnutrition will be provided to both groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- (i) ONS + Exercise group (Experimental): This group will consume whey protein ONS enriched with leucine and vitamin D, twice a day for 12 weeks. The optimal time to consume the ONS on non-exercise days will be based on each participants 24-hour dietary recall. On exercise days, participants will be asked to consume the ONS after breakfast and after the exercise class. Participants will participate in a resistance-based exercise programme twice a week for 12 weeks which will be carried out over Zoom. Standard dietary advice to increase intake of protein, leucine and vitamin D using available literature designed for those at risk of malnutrition will be provided to this group by the research nutritionist.
  Interventions: Dietary Supplement: Fortimel Advanced, Nutricia; Other: Resistance Exercise programme; Other: Dietary advice
- (ii) Exercise-alone group (Active Comparator): Participants will participate in a resistance-based exercise programme twice a week for 12 weeks which will be carried out over Zoom. Standard dietary advice to increase intake of protein, leucine and vitamin D using available literature designed for those at risk of malnutrition will be provided to this group by the research nutritionist. The participants will not be provided with a placebo ONS.
  Interventions: Other: Resistance Exercise programme; Other: Dietary advice

INTERVENTIONS:
Dietary Supplement: Fortimel Advanced, Nutricia — Per 200 mL serving size: 300 kcal, 21 g whey protein, 3 g leucine & 10 µg Vitamin D.
  Arms: (i) ONS + Exercise group
Other: Resistance Exercise programme — Participants will participate in the resistance-based exercise programme twice a week for 12-weeks via Zoom. Each session will last between 45-60 minutes with 2-3 sets and 8-12 reps, twice a week for the 12 weeks.
Other: Dietary advice — Standard dietary advice to increase intake of protein, leucine and vitamin D using available literature designed for those at risk of malnutrition will be provided to both groups by the research nutritionist. Literature provided will include booklets containing lists of foods high in protein, leucine and vitamin D plus easy-to-prepare meal ideas. The dietary advice provided will be informed by the 24-hour dietary recall information obtained from each participant.

SUMMARY:
To explore the effectiveness of a 12-week resistance exercise programme plus or minus an oral nutritional supplement on the nutritional status of community-dwelling older adults who receive home care and are at risk of sarcopenia.

DETAILED DESCRIPTION:
The aim of this study is to investigate the effectiveness of consuming a whey-based protein ONS enriched with leucine and vitamin D, in conjunction with an online resistance-based exercise programme, versus the effectiveness of an online exercise programme alone, for twelve weeks, in a cohort of older adults who are at risk of sarcopenia and who require supportive home care.

The primary outcome will be functional and nutritional status measured using the Timed get Up and Go (TUG) test and the full form of the mini-nutritional assessment (MNA-FF). The secondary outcomes include feasibility of implementation, defined by recruitment, retention and adherence rates, measures of body composition, muscle strength and quality of life.

The groups will be as follows: (i) whey protein ONS enriched with leucine and vitamin D plus an online exercise programme or (ii) an online exercise programme alone.

The exercise programme will be comprised of two sessions per week for 12-weeks and will be delivered using the UCD Zoom platform. The exercise programme will include strength movements that are intended to build muscle mass and improve physical function. The exercise programme will involve four phases split over the 12-week intervention: phase 1 (2 weeks), phase 2 (3 weeks), phase 3 (3 weeks) and phase 4 (4 weeks).

The ONS is a high protein, leucine and vitamin D enriched drink. Participants randomised to the ONS group will be asked to consume the drink twice a day for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Older adults (70+ years)
* Requiring supportive homecare
* At risk of sarcopenia

Exclusion Criteria:

* Cognitive impairment
* Severe kidney disease (glomerular filtration rate < 30 mL/min)
* Moderate to severe liver disease (Child-Pugh class B or C)
* Psychiatric disorder
* Receiving treatment or palliative care for cancer
* Receiving enteral or parenteral nutrition
* Hypersensitivity to any component of ONS
* Taking ONS
* Allergic to dairy products
* Regularly undertaking resistance (strength) training
* Advised by GP not to undertake physical activity

Ages: 70 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline functional status at 12 weeks | 12 weeks
  Timed Get Up & Go test will be used to assess physical performance as advised by the EWGSOP2 to test for sarcopenia.
Change from baseline nutritional status at 12 weeks | 12 weeks
  The nutritional status of participants will be assessed using the full form of the mini-nutritional assessment-full form (MNA-FF). 24 - 30 points indicates normal nutrition status; 17 to 23.5 points indicates at risk of malnutrition & less than 17 points indicates malnutrition.

SECONDARY OUTCOMES:
Adherence | 12 weeks
  Attendance at the resistance exercise classes + consumption of the protein supplement
Muscle mass | Values at baseline will be compared to values recorded at 12 and at 24 weeks
  Muscle mass will be assessed using Bioelectrical Impedance Analysis
Muscle strength | Values at baseline will be compared to values recorded at 12 and at 24 weeks
  Handgrip strength will be used to assess upper-body strength
Five Times Sit-To-Stand test | Values at baseline will be compared to values recorded at 12 and at 24 weeks
  Five Times Sit-To-Stand test will be used to assess lower extremity strength
4 m Gait Speed test | Values at baseline will be compared to values recorded at 12 and at 24 weeks
  4 m Gait Speed test will be used to assess physical performance as advised by the EWGSOP2 to test for sarcopenia
Change in self-reported quality of life | Values at baseline will be compared to values recorded at 12 and at 24 weeks
  The Health Related Quality of Life 12-Item Short Form Survey (SF-12v2) will be used to assess participants quality of life. Score ranges from 0 - 100, higher score indicates higher quality of life.
Change in risk of depression | Values at baseline will be compared to values recorded at 12 and at 24 weeks
  The Geriatric Depression Score-15 item questionnaire will be used to screen for risk of depression in the participants. Score of 0-5 is normal & score greater than 5 suggests risk of depression.
Change in functional status | Values at baseline will be compared to values recorded at 12 and at 24 weeks
  The Katz Index of Independence in Activities of Daily Living will be used to assess functional status. Score of 6 indicates full function, 4 indicates moderate impairment, and 2 or less indicates severe functional impairment.
Change in baseline nutritional status at week 24 | 24 weeks
  The nutritional status of participants will assessed using the full form of the mini-nutritional assessment-full form (MNA-FF). 24 - 30 points indicates normal nutrition status, 17 to 23.5 points indicates at risk of malnutrition & less than 17 points indicates malnutrition.
Change from baseline functional status at 24 weeks | 24 weeks
  Timed Get Up & Go test will be used to assess physical performance as advised by the EWGSOP2 to test for sarcopenia.
Retention | Up to 24 weeks
  The number of participants retained at the end of the study
Recruitment | Up to 24 weeks
  The number of participants recruited divided by the number of eligible participants.

CONTACTS AND LOCATIONS:
Locations (1):
- UCD School of Public Health, Physiotherapy and Sports Science, Dublin, Leinster, Ireland

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.

REFERENCES:
- [Derived] Fallon CM, Cunningham CG, Horner K, Corish CA. Oral nutritional supplement combined with an online resistance training programme to improve physical function and nutritional status in older adults receiving home care and at risk of sarcopenia: protocol for the randomised controlled POWER trial. HRB Open Res. 2026 Jan 20;8:41. doi: 10.12688/hrbopenres.14086.3. eCollection 2025. PMID 41467085